CLINICAL TRIAL: NCT03126604
Title: Evaluation of Pelvic Floor Function After Vaginal and Cesarean Delivery Among Egyptian Women
Brief Title: Pelvic Floor Function After Vaginal and Cesarean Delivery Among Egyptian Women
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Professor, Cairo University
Other Study IDs: 5
Record Dates: First submitted 2017-04-20; First posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Pelvic Floor Disorders
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- vaginal delivery: Women underwent non complicated non instumental normal vaginal delivery
  Interventions: Diagnostic Test: female sexual function index
- Cesarean section: Women underwent elective Cesarean section
  Interventions: Diagnostic Test: female sexual function index

INTERVENTIONS:
Diagnostic Test: female sexual function index — evaluation of sexual functions questionnaire about Desire, Arousal, Orgasm,pain , lubrications, satisfactions

SUMMARY:
A cross sectional study for assessment of pelvic floor functions after 6 months to 4 years after normal vaginal delivery or Cesarean section

DETAILED DESCRIPTION:
A cross sectional study for assessment of pelvic floor functions after 6 months to 4 years after normal vaginal delivery or Cesarean section Four separate entities were evaluated using internationally recognized and validated questionnaires:

1. Pelvic organ prolapse evaluated using the Pelvic Organ Prolapse Distress Inventory
2. Urinary functions were evaluated using the International Consultation on Incontinence Questionnaire Short Form
3. Fecal incontinence was evaluated using Wexner Fecal Incontinence Score
4. Sexual functions were evaluated using female sexual function index

ELIGIBILITY:
Inclusion Criteria:

* primiparity,
* singleton pregnancy
* cephalic presentation
* term delivery (38-42 weeks).

Exclusion Criteria:

* Women with operative vaginal delivery (vacuum extraction or forceps delivery)
* women who had another delivery between the time of first one and time of evaluation
* women with neurological diseases
* women with vascular diseases and Diabetes Mellitus

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: women who delivered vaginally or Cesarean for the first time within 6 months to 5 years before evaluation
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
urinary incontinence | 6 months after delivery
  evaluation using the International Consultation on Incontinence Questionnaire Short Form

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes